CLINICAL TRIAL: NCT03461380
Title: Efficacy of Menopause Relief EP-40 - Fixed Combination of Cimicifuga EP-40 and Rhodiola EPR-7 Extracts in Women With Menopausal Symptoms: A Randomized, Double Blind, Placebo Controlled Study
Brief Title: Effect of Menopause Relief EP-40 in Women With Menopausal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EuroPharma, Inc. (Industry)
Collaborators: I.Zhordania Institute of Reproductology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EP-1002; EP-2018-1 (Other: Sponsor)
Record Dates: First submitted 2018-03-02; First posted 2018-03-12 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Menopause
Keywords: Cimicifuga, Rhodiola, Menopause Symptoms
MeSH Terms: interventions — black cohosh root extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Menopause Relief EP-40 (Experimental): Fixed combination of black cohosh EP-40 and Rhodiola rosea EPR-7 206.5 mg orally twice daily; daily dose 413 mg of active ingredients
  Interventions: Dietary Supplement: Menopause Relief EP-40
- High Dose Black Cohosh (Active Comparator): Black cohosh 500 mg orally twice daily; daily dose 1000 mg of active ingredient
  Interventions: Dietary Supplement: High Dose Black Cohosh
- Placebo (Placebo Comparator): Placebo capsule 600 mg excipients orally twice daily
  Interventions: Dietary Supplement: Placebo
- Low Dose Black Cohosh (Active Comparator): Black cohosh 6.5 mg orally twice daily; daily dose 13 mg of active ingredient
  Interventions: Dietary Supplement: Low Dose Black Cohosh

INTERVENTIONS:
Dietary Supplement: Menopause Relief EP-40 — Fixed combination of black cohosh and Rhodiola rosea
  Arms: Menopause Relief EP-40
Dietary Supplement: Low Dose Black Cohosh — 6.5 mg black cohosh
  Arms: Low Dose Black Cohosh
Dietary Supplement: High Dose Black Cohosh — 500 mg black cohosh
  Arms: High Dose Black Cohosh
Dietary Supplement: Placebo — 600 mg excipient
  Arms: Placebo

SUMMARY:
This study compares the efficacy of a fixed combination of black cohosh (EP-40) and Rhodiola rosea (EPR-7) with low (6.5 mg) and high doses (500 mg) of a standardized black cohosh extract only in adult woman with menopausal complaints.

DETAILED DESCRIPTION:
Due to the problems caused by Hormone Replacement Therapy with chemical entities, some medicinal plants used in the traditional systems of medicine have shown immense potential in non-hormonal treatment of menopausal symptoms without major adverse events. We hypothesize that Menopause Relief EP-40 (a fixed combination of Cimicifuga EP-40 and Rhodiola EPR-7 extracts) will significantly relieve menopausal complaints such as hot flushes, profuse sweating hot flushes, excessive perspiration, night sweats, sleep disorders, nervousness, mood swings, physical and mental fatigue as compared to EP-40® capsules or placebo in adult females in menopause.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of menopausal female climacteric states (N95.1 according to the International Statistical Classification of Diseases and Related Health Problems 10th Revision, ICD-10, Version for 2014) which is characterized by symptoms such as flushing, sleeplessness, headache, lack of concentration associated with menopause, etc
* Patients suffering from menopausal syndrome with neurovegetative components which have been stable anamnestically during the last 2 weeks
* No medication taken for management of menopausal syndrome with neurovegetative components during the last 4 weeks
* Ability to understand and provide signed informed consent
* Ability to participate in the study
* In some cases, diagnosis should be confirmed by blood tests of follicle-stimulating hormone (≥ 40 IU/L) [postmenopausal status], thyroid function with normal serum free T4 (fT4), estrogen (estrodiol levels) [premenopausal 30-400 pg/mL; after menopause <30 pg/mL]

Exclusion Criteria:

* subjects with previous or current psychological disease that could interfere with their ability to participate in the study
* anamnestic or current alcohol or drug abuse
* concomitant treatment with psychotropic (in particular benzodiazepines, antidepressants, hypnotics or neuroleptics, tamoxifen, clomiphene, and danazol) or hormonally acting drugs such as hormone replacement therapy (HRT)
* hyperthyroidism
* malignant tumors
* continuous climacteric bleeding and complaints related to myomas
* patients who have taken another experimental drug within a 4-week period prior to the trial
* pregnancy/lactation
* serious internal disease
* previous organ transplantation
* premenopausal women with insufficient contraceptive protection
* hypersensitivity to one of the ingredients of the trial medication
* a body mass index of >30

Min Age: 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Kupperman Menopausal Index (KMI) | 12 weeks
  A modified total Kupperman Index (KMI) score and its sub-items will be used. It is a 10-item questionnaire of single symptoms with scores ranging from 0 to 3 (none, mild, moderate and severe). Total KMI is defined as the sum of sub-item scores multiplied by any weighting factors. The maximum value of the total KMI is 48. The primary outcome will be the difference in the changes from baseline to the end of therapy (week 12), between verum groups and placebo, assessed by the total KMI and stratified by individual baseline scores in an intention-to-treat (ITT) analysis (patients treated with study medication and with at least one efficacy assessment after baseline).
Menopause Rating Scale (MRS) | 12 weeks
  The MRS is a patient reported assessment of 11 symptoms of menopause on a scale of 0 (none) to 4 (very severe). The MRS groups symptoms into three subscales: psychological, somatic, and urogenital. A composite score is calculated by adding the items in each dimension (subscale). The total score is the sum of the three dimensional scores. The primary outcome will be the difference in the changes from baseline to the end of therapy (week 12), between both verum groups and placebo, assessed by the MRS and stratified by individual baseline scores in an intention-to-treat (ITT) analysis (patients treated with study medication and with at least one efficacy assessment after baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Lali Phkhaladze, PhD, MD, Principal Investigator — I.Zhordania Institute of Reproductology, Tevdore Mgvdeli Street, Tbilisi, Georgia
Locations (1):
- I.Zhordania Institute of Reproductology, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No